CLINICAL TRIAL: NCT02053324
Title: A Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, Dosimetry, Maximum Tolerated Dose and Preliminary Efficacy of Intra-lesionally Injected AvidinOX, Followed by Systemic IV Administration of Escalating Doses of [177Lu]DOTA-biotin in Patients With Liver Metastases From Colorectal Cancer
Brief Title: AvidinOX + [177Lu]DOTA-biotin (or 177Lu-ST2210) Complex in Patients With Liver Metastases From Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AvOX/ST2210-CR-12-001; 2012-005577-32 (EudraCT Number)
Record Dates: First submitted 2014-01-24; First posted 2014-02-03 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Liver Metastases
Keywords: AvidinOX

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation design
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AvidinOX/ST2210 (Experimental): AvidinOX/ST2210 - vial containing 22.5 mg AvidinOX + vials containing 10 ml of water for injection (WFI) for the reconstitution in a clear solution with an AvidinOX concentration of 3 mg/ml. One Intralesion administration of a volume of reconstituted AvidinOX equal to 15 % of the lesion volume followed by intravenous infusion of 177Lu-ST2210 Diagnostic dose : 10 ml, 250 MBq±10%177Lu, approximately 1 mg ST2210, 100 mg/mL ascorbic acid, followed by intravenous infusion of a therapeutic dose: 25 ml, escalating 177Lu dose starting at 5 Gigabequerel (GBq) ±10%with escalation steps of 2.5 GBq up to 15 GBq ±10%, approximately 1 mg ST2210, 100 mg/ml ascorbic acid
  Interventions: Combination Product: AvidinOX/ST2210

INTERVENTIONS:
Combination Product: AvidinOX/ST2210 — One intralesion injection of AvidinOX followed by an intravenous infusion of ST2210

SUMMARY:
The purpose of the study is to assess a new treatment for patients with liver tumor metastases from colorectal cancer. The treatment has never been used in humans before. The treatment foresees the use of two compounds: AvdinOX and [177Lu]DOTA-biotin.

AvidinOX is a new compound, essentially a natural protein obtained from hen eggs, while [177Lu]DOTA-biotin is a new chemical compound resulting from the combination of the DOTA-biotin (also deriving from a natural vitamin which is biotin) with the 177Lutetium, an atom which emits radiation.

AvidinOX will be injected directly into the metastases in the liver and [177Lu]DOTA-biotin will be injected into the arm vein.

One specific property of AvidinOX is that it chemically links to the tumor tissues when it is injected while maintaining the capacity to take up [177Lu]DOTA-biotin. Once locally bound in tumor tissue, AvidinOX becomes an "artificial receptor" for intravenously injected [177Lu]DOTA-biotin, which allows an internal radiation therapy of the tumor tissue.

The treatment of liver metastases with local injection of AvidinOX and the following intra-venous injection of [177Lu]DOTA-biotin could be simpler and more tolerable than the current available treatments.

DETAILED DESCRIPTION:
Primary objectives

1. To identify the Maximum Tolerated Dose (MTD) of 177Lu-ST2210 after prior intra-lesional injection of AvidinOX in the liver.
2. To assess safety and tolerability of intra-lesionally injected AvidinOX + IV injected 177Lu-ST2210
3. To evaluate intra-lesional distribution and retention of AvidinOX + 177Lu-ST2210 complex in liver metastases
4. To evaluate systemic biodistribution and pharmacokinetics of 177Lu-ST2210 and {AvidinOX + 177Lu-ST2210}- complex

Secondary objectives

1. To evaluate proportional 177Lu-ST2210 tumor binding, as a function of total tumor load, and AvidinOX dose injected
2. To demonstrate AvidinOX post-deposition reactivity with 177Lu-ST2210 over time
3. To evaluate whole body dosimetry of IV 177Lu-ST2210 after prior AvidinOX injection (radiation safety dosimetry)
4. To record individual tumor dosimetry
5. To evaluate preliminary efficacy of {AvidinOX + 177Lu-ST2210}-complex in reducing tumor size
6. To evaluate whole body safety dosimetry and dose linearity of IV administered 177Lu-ST2210 after prior intra-lesional injection of AvidinOX
7. To evaluate pharmacokinetics of ST2210 in plasma and urine

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Liver metastases from histologically confirmed colorectal cancer and at least one liver metastasis ≥ 1 cm (measurable disease), which is chemo-resistant, not eligible for curative surgery and suitable for intra-lesional injection as assessed by the investigator.
3. Total liver tumor burden requiring ≤ 75 ml AvidinOX
4. Maximum of 9 liver metastases
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
6. Life expectancy of at least 3 months.
7. Clotting parameters as follows, with local normal ranges to be taken as reference:

   * Prothrombin Time (Quick).Patients showing an increase of the Upper Limit of the Normal (ULN) range of about 20% can also be considered for inclusion.
   * International Normalised Ratio (INR). Patients showing an increase of the ULN of about 20% can also be considered for inclusion
   * Activated Partial Thromboplastin Time (aPTT). Patients showing an increase of the ULN of about 20% can also be considered for inclusion
   * Fibrinogen. Patients showing a decrease of the Lower Limit of the Normal range (LLN) of about 20% can also be considered for inclusion.
8. Haematological, liver and renal function test results ≤ grade 2 toxicity (according to US National Cancer Institute's "Common Terminology Criteria for Adverse Events v4.03 [CTCAE]"), i.e.:

   * Haematology:

     * Haemoglobin ≥ 8 g/dl
     * White blood cell count ≥ 2 x 109/L
     * Platelets ≥ 80x 109/L
   * Liver:

     * Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (AP) ≤ 5 times upper limit of normal
     * Bilirubin ≤ 3 times upper limit of normal
   * Renal:

     * Urine protein dipstick: 0
     * estimated Glomerular Filtration Rate (eGFR)> 30 ml/min/1.73 m2 (with CKD-EPI formula)
9. Written informed consent

Exclusion Criteria:

1. Known hypersensitivity to Avidin or AvidinOX (e.g. hen egg)
2. Known hypersensitivity to ST2210(DOTA biotin) or any excipient.
3. Life limiting metastases outside the liver. Metastases outside the liver are allowed only in case the residual metastases (after liver treatment) are amenable to further treatments (e.g. surgical removal)
4. Presence of unreachable (e.g. located in a region in the liver that cannot be reached by needle, or too close to major blood vessels or adjacent to main organs) or untreatable hepatic lesions so that the benefit from the treatment of the treatable lesions does not justify patient's inclusion
5. Active infection at screening or history of severe infection within the previous 3 months, if clinically relevant at screening as considered by the investigator
6. Known human immunodeficiency virus (HIV) positive serology or chronically active hepatitis B or C.
7. Administration of another investigational medicinal product within 30 days before the screening period.
8. Previous treatment with Selective Internal Radiation Therapy (SIRT) spheres or any radiopharmaceutical within a period corresponding to 8 half-lives of the radionuclide used for labeling the respective radiopharmaceutical prior to the administration of study drug.
9. Women of child-bearing potential. A permanent postmenopausal status must be proven as follows: history of hysterectomy or hormone analysis in serum: estradiol < 20 pg/ml and follicle stimulating hormone (FSH) > 40 IU/L, or amenorrhea starting at least 1 year prior to the study start andnegativeβHCG .
10. Men unwilling to use appropriate contraceptive methods during the study and up to six months after the end of the study
11. Inability or unwillingness to be catheterized
12. History of somatic or psychiatric disease/condition that may interfere with the objectives of the study
13. Clinically significant illness or clinically relevant trauma within 15 days before the screening period
14. Patient who underwent chemotherapy, radiation therapy within 15 days before the screening period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity evaluated using NCI Common Toxicity Criteria (CTCAE 4.03) | up to six weeks

SECONDARY OUTCOMES:
Adverse Events | up to 1 year

OTHER OUTCOMES:
tumor response | 1 year
  Tumor response according to Response Evaluation Criteria in Solid Tumors (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Haug, MD, Principal Investigator — Allgemeines Krankenhaus Wien (Austria); Andreas Wicki, MD, Principal Investigator — Universitatsspital Basel (Switzerland); Francesco Scopinaro, MD, Principal Investigator — St. Andrea Hospital Rome (Italy); Roberto Cianni, MD, Principal Investigator — S Maria Goretti Hospital - Latina (Italy); Michele Sicolo, MD, Principal Investigator — Dell'Angelo Hospital - Mestre (Italy)
Locations (4):
- Allgemeines Krankenhaus Wien, Vienna, Austria
- Italy (3):
  - Ospedale S. Maria Goretti, Latina, ROME
  - Ospedale dell' Angelo di Mestre, Mestre, Venice
  - S. Andrea Hospital, Rome

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vesci L, Carollo V, Rosi A, De Santis R. Therapeutic efficacy of intra-tumor AvidinOX and low systemic dose biotinylated cetuximab, with and without cisplatin, in an orthotopic model of head and neck cancer. Oncol Lett. 2019 Mar;17(3):3529-3536. doi: 10.3892/ol.2019.10003. Epub 2019 Feb 1. PMID 30867794
- [Derived] Milazzo FM, Anastasi AM, Chiapparino C, Rosi A, Leoni B, Vesci L, Petronzelli F, De Santis R. AvidinOX-anchored biotinylated trastuzumab and pertuzumab induce down-modulation of ErbB2 and tumor cell death at concentrations order of magnitude lower than not-anchored antibodies. Oncotarget. 2017 Apr 4;8(14):22590-22605. doi: 10.18632/oncotarget.15145. PMID 28186982
- [Derived] Vesci L, Milazzo FM, Anastasi AM, Petronzelli F, Chiapparino C, Carollo V, Roscilli G, Marra E, Luberto L, Aurisicchio L, Pacello ML, Spagnoli LG, De Santis R. Intra-tumor AvidinOX allows efficacy of low dose systemic biotinylated Cetuximab in a model of head and neck cancer. Oncotarget. 2016 Jan 5;7(1):914-28. doi: 10.18632/oncotarget.6089. PMID 26575422
- [Derived] Albertoni C, Leoni B, Rosi A, D'Alessio V, Carollo V, Spagnoli LG, van Echteld C, De Santis R. Radionuclide Therapy of Unresectable Tumors with AvidinOX and (90)Y-biotinDOTA: Tongue Cancer Paradigm. Cancer Biother Radiopharm. 2015 Sep;30(7):291-8. doi: 10.1089/cbr.2015.1837. Epub 2015 Jul 13. PMID 26167947